CLINICAL TRIAL: NCT00278577
Title: Immune Ablation and Hematopoietic Stem Cell Support in Patients With Severe Crohn's Disease
Brief Title: Hematopoietic Stem Cell Support in Patients With Severe Crohn's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Richard Burt, MD (Other)
Responsible Party: Sponsor-Investigator, Richard Burt, MD, MD, Northwestern University
Organization: Northwestern University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 97CD1; NCT00014703 (obsolete NCT alias)
Record Dates: First submitted 2006-01-15; First posted 2006-01-18 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-04

CONDITIONS: CROHN'S DISEASE
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Hematopoietic Stem Cell Transplant (Experimental)
  Interventions: Biological: Immune Ablation and Hematopoietic Stem Cell Support

INTERVENTIONS:
Biological: Immune Ablation and Hematopoietic Stem Cell Support — Autologous Hematopoietic Stem Cell Transplant

SUMMARY:
This disease is believed to be caused by immune cells (called lymphocytes) attacking tissue. Risk of death is highest in people with active acute disease. In addition, progressive Crohn's Disease leads to further loss of bowel function, which may eventually result in the need for artificial nutritional support (parenteral nutrition).

This study involves high dose chemotherapy followed by return (infusion) of blood stem cells. Stem cells are undeveloped cells that have the capacity to grow into mature blood cells, which normally circulate in the blood stream. The high dose chemotherapy consists of cyclophosphamide and anti lymphocyte antibody (a protein that depletes cells that cause damage to the body). The purpose of the intense chemotherapy is to destroy the immune system completely. The purpose of the stem cell infusion is to restore the body's blood production, which will be severely impaired by the high dose chemotherapy and anti lymphocyte antibody.

ELIGIBILITY:
Inclusion Criteria:

1. Less than physiologic age 60 at time of pretransplant evaluation
2. An established clinical diagnosis of severe CD that has failed therapy with prednisone, azathioprine, 5 ASA products and metronidazole, and has failed an anti-TNF alpha inhibitor. Failure is defined as a CDAI (appendix A) 250-400 or a Craig Severity Score that is > 17 (appendix D)
3. Pre-study peripheral blood counts must include a platelet count greater than 100,000/ul and an absolute neutrophil count greater than 1500/ul.
4. Stem cell harvest greater than 1.4 x 106 CD34 cells/kg after CD34+ selection (to continue to transplant)
5. Ability to give informed consent

Exclusion Criteria

1. HIV positive
2. History of coronary artery disease, or congestive heart failure
3. Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemotherapy
4. Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as head and neck cancer, or stage I breast cancer will be considered on an individual basis
5. Positive pregnancy test, lactation, inability or unwillingness to pursue effective means of birth control, failure to accept or comprehend irreversible sterility as a side effect of therapy
6. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible
7. FEV I/FVC < 50% of predicted, DLCO < 50% of predicted
8. Resting LVEF < 40%
9. Bilirubin > 2.0 mg/dl, transferase (AST) > 2x upper limit of normal, unless the abnormalities are secondary to Crohn's disease
10. Serum creatinine > 2.0 mg/dl
11. Platelet count less than 100,000/ul, ANC less than 1500/ul
12. Patients presenting with intestinal perforation or toxic megacolon, or a suppurative problem that will require urgent surgery. In addition, the patient may not have any active infection. The presence of intestinal stomas does not exclude the patient from study.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2001-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
11.1 CDAI - If the index worsens by 50 points for more than 4 weeks, the disease will be considered progressive; if it improves by 70 points for more than four weeks, it will be considered improved; otherwise it will be considered stable. | 5 years after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Robert Craig, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States